CLINICAL TRIAL: NCT05872048
Title: Assessment of Orthodontic Canine Retraction Via Two Approaches of Periodontal Distraction: A Comparative Clinical Study
Brief Title: Evaluation of Periodontal Distractor in Acceleration of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Mohamed El-Hendawey, Assistant lecturer, Deparement of Orthodontics, Al Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: distraction in orthodontics
Record Dates: First submitted 2023-03-07; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Canine Retraction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periodontal distractor with interseptal bone cuts (Experimental)
  Interventions: Device: periodontal distractor
- periodontal distractor without interseptal bone cuts (Experimental)
  Interventions: Device: periodontal distractor

INTERVENTIONS:
Device: periodontal distractor — custom made device from hyrex screw

SUMMARY:
evaluate the effect of periodontal distractor with and without interseptal bone cuts on the displacement of the maxillary canines, to assess the effect of two approaches on the pain intensity and on the pulp vitality of the retracted canines.

DETAILED DESCRIPTION:
The sample of the study consisted of 32 canines in 16 female patients (16- 21 years old) requiring extraction of bilateral maxillary first premolars and canine retraction. They were divided into two groups: canine retraction was done by buccal periodontal distractor with distal interseptal bone cuts (Group I), canine retraction was done by buccal periodontal distractor without distal interseptal bone cuts (Group II). After bilateral maxillary premolar extraction in both groups inter septal bone cuts was done in group I only. Then the periodontal distractor was cemented and activated twice per day in both groups. Rate of canine retraction was evaluated before and after complete canine retraction direct in patient's mouth with digital caliper. Pain intensity was evaluated at 1st ,2nd ,4th and 7th days after activation through visual analog scale (VAS). An electrical vitality test was evaluated before and after the distraction procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: 16-21 years.
* patients required bilateral extraction of maxillary first premolars followed by maxillary canine retraction (class I malocclusion as excessive overjet, bimaxillary protrusion, class II malocclusion).
* The dentition didn't exhibit any gross anatomic root anomalies as assessed from panoramic radiographs.
* No systemic disease that may affects the bone.
* No periodontal disease.
* Good oral hygiene.
* Very good patient compliance.
* Absence of any previous orthodontic treatment.

Exclusion Criteria:

* The dentition exhibit any gross anatomic root anomalies as assessed from panoramic radiographs.
* Cases with deep carious lesions or endodontic lesions involving the maxillary canines and buccal segments.
* Cases with severly rotated or grossly malpositioned canines.
* Systemic disease that may affects the bone.
* Periodontal disease and poor oral hygiene.
* Presence of previous orthodontic treatment.

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
rate of canine retraction | one month
  amount of distalization\time

SECONDARY OUTCOMES:
pain intensity | one month
  visual analog scale minimum score = 0 maximum score = 10 higher scores mean worse outcome

OTHER OUTCOMES:
pulp vitality | two months
  electric pulp tester

CONTACTS AND LOCATIONS:
Overall Officials: Maha M Mohamed, assistant professor, Study Director — Assistant professor of orthodontics, Faculty of Dental Medicine, Al Azhar Univeristy, Cairo; Farouk A Hussein, Professor, Study Chair — professor of orthodontics, Faculty of Dental Medicine, Al Azhar Univeristy, Cairo; Suzan A Hssan, professor, Study Chair — professor of oral sugery, Faculty of Dental Medicine, Al Azhar Univeristy, Cairo
Locations (1):
- Faculty of Dental Medicine, Al Azhar University, Cairo, Egypt